CLINICAL TRIAL: NCT00258960
Title: Phase IV/II Trial With the Combination of Pegylated Liposomal Doxorubicin (Caelyx), Cyclophosphamide and Trastuzumab in Patients With Metastatic Breast Cancer With Overexpression of Human Epidermal Growth Factor Receptor 2 (HER2)/Neu
Brief Title: Caelyx, Cyclophosphamide and Herceptin in Patients With Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Spanish Breast Cancer Research Group (Other)
Collaborators: Schering-Plough (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GEICAM/2004-05
Record Dates: First submitted 2005-11-24; First posted 2005-11-28 (Estimated); Results first posted 2019-07-15 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-04

CONDITIONS: Breast Cancer
Keywords: HER2 positive breast cancer; Metastatic breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — liposomal doxorubicin; Cyclophosphamide; Trastuzumab

ARMS (1):
- Caelyx,Cyclophosphamide,Trastuzumab (Other): Caelyx (Liposomal Doxorubicin) 50 mg/m2 every 4 weeks for 6 cycles, Cyclophosphamide 600 mg/m2 every 4 weeks for 6 cycles, Trastuzumab weekly for 24 weeks, at dose of 2mg/kg (day 1 loading dose of 4mg/kg)
  Interventions: Drug: Liposomal Doxorubicin; Drug: Cyclophosphamide; Drug: Trastuzumab

INTERVENTIONS:
Drug: Liposomal Doxorubicin
  Other Names: Caelyx
Drug: Cyclophosphamide
  Other Names: Cytoxan
Drug: Trastuzumab
  Other Names: Herceptin

SUMMARY:
Eligible patients must receive Caelyx plus Cyclophosphamide plus Herceptin for 6 cycles that will be administered every 4 weeks.

DETAILED DESCRIPTION:
Sample size calculation will be done by means of Simon's method in 2 stages for phase II studies and will be based on the principal aim of the study (evaluation of the rate of objective response).

The hypothesis brings over of the efficiency of the treatment it will be accepted if a rate of objective response of at least 55 % is obtained, rejecting the efficiency of the treatment when the rate of response targets be lower than 35 %. In this case, considering an alpha error of 0.05 and 80 % power, 14 patients will be included in the first stage; the study would continue if more than 5 objective responses were found. The total number of patients to including in the study would be 44. The results will be significant if they find at least 20 objective responses.

Assuming a drop-out rate of 10 %, the total number of patients needed is 49 patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients must sign an informed consent before of specific procedures of clinical trial.
* Patients with histologically confirmed breast cancer and overexpression of Her2neu.
* Age> 18 years.
* Eastern Cooperative Oncology Group (ECOG) equal or < 2.
* Patients have not been treated previously with chemotherapy for metastatic disease.
* Patients must have at least one measurable lesion according to RECIST criteria.
* Patients should have an adequate organ function to tolerate chemotherapy.

Exclusion Criteria:

* Patients with hypersensitivity reactions to any of the medications of the clinical trial.
* Patients who are pregnant or lactating are not eligible.
* Hepatic disease.
* Not controlled active infection
* Symptomatic metastatic brain cancer
* Previous adjuvant treatment with anthracyclines with a total accumulated dose > 300 mg/m2 (Doxorubicin) or > 600 mg/m2 (Epirubicin)

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2006-02-15 (Actual); Primary Completion 2008-07 (Actual); Study Completion 2009-07-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Hospital Clínico Universitario San Carlos
Locations (12):
- Spain (12):
  - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Fundación Hospital Alcorcón, Alcorcón, Madrid
  - Hospital Juan Canalejo, A Coruña
  - Centro Oncológico Regional de Galicia, A Coruña
  - Hospital Clinic i Provincial, Barcelona
  - Hospital Puerta del Mar, Cadiz
  - Hospital Provincial de Castellón, Castelló
  - Complejo Hospitalario de Jaen, Jaén
  - Hospital Xeral Calde de Lugo, Lugo
  - Hospital Universitario Doce de Octubre, Madrid
  - Hospital Clínico Universitario San Carlos, Madrid
  - Hospital Nuestra Señora de Candelaria, Santa Cruz de Tenerife

REFERENCES:
- [Result] Martin M, Sanchez-Rovira P, Munoz M, Baena-Canada JM, Mel JR, Margeli M, Ramos M, Martinez E, Garcia-Saenz JA, Casado A, Jaen AM, Gonzalez-Farre X, Escudero MJ, Rodriguez-Martin C, Carrasco E; GEICAM. Pegylated liposomal doxorubicin in combination with cyclophosphamide and trastuzumab in HER2-positive metastatic breast cancer patients: efficacy and cardiac safety from the GEICAM/2004-05 study. Ann Oncol. 2011 Dec;22(12):2591-2596. doi: 10.1093/annonc/mdr024. Epub 2011 Mar 17. PMID 21421542
- See also: Spanish Breast Cancer Research Group (GEICAM) is a Spanish Breast Cancer Research Group — http://www.geicam.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between February 2006 and June 2008, 49 patients were enrolled at 12 Spanish sites. One patient never received treatment due to early death from progressive disease and was not included in this analysis.
Groups:
- Liposomal Doxorubicin,Cyclophosphamide,Trastuzumab: Liposomal Doxorubicin 50 mg/m2 every 4 weeks for six cycles, Cyclophosphamide 600 mg/m2 every 4 weeks for six cycles, Trastuzumab weekly for 24 weeks, at dose of 2mg/kg (day 1 loading dose of 4mg/kg)
  Liposomal Doxorubicin
  Cyclophosphamide
  Trastuzumab
Period: Overall Study
Arm/Group | Liposomal Doxorubicin,Cyclophosphamide,Trastuzumab
Started | 49 (49 patients included but 1 is not considered due to not receive any treatment and died before start)
Completed | 32
Not Completed | 17
Not completed — Death | 2
Not completed — Disease Progression | 7
Not completed — Adverse Event | 4
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 1
Not completed — Mistake | 2

BASELINE CHARACTERISTICS:
Population: Between February 2006 and June 2008, 49 patients were enrolled at 12 Spanish sites. One patient never received treatment due to early death from progressive disease and was not included in this analysis.
Arm/Group | Liposomal Doxorubicin,Cyclophosphamide,Trastuzumab
Number analyzed (Participants) | 48
Age, Continuous [Median (Full Range); unit: years] — Patient included by error at 78 years.
  years | 57 [37 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48
  Male | 0
Eastern Cooperative Oncology Group (ECOG) [Count of Participants; unit: Participants] — Measure Description: ECOG score runs from 0 to 5, with 0 denoting perfect health and 5 death.
  0 - Asymptomatic
  1. - Symptomatic but completely ambulatory
  2. - Symptomatic, <50% in bed during the day
  3. - Symptomatic, >50% in bed, but not bedbound
  4. - Bedbound
  5. - Death
  Participants
    ECOG 0 | 26
    ECOG 1 | 20
    ECOG 2 | 2
Menopausal Status [Count of Participants; unit: Participants]
  Premenopausal | 9
  Postmenopausal | 39
Hormonal receptor status [Count of Participants; unit: Participants] — A cancer is called hormonal receptor positive if it has receptors for progesterone or estrogen. This suggests that the cancer cells, like normal breast cells, may receive signals from progesterone or estrogen that could promote their growth.
  If the cancer is hormone-receptor-negative (no receptors are present), then hormonal therapy is unlikely to work.
  Participants
    Positive | 24
    Negative | 24
Disease stage at diagnosis [Count of Participants; unit: Participants] — TNM staging system:
  Stage (S) 0: noninvasive ductal carcinoma in situ S IA: tumor small, invasive S IB: spread to the lymph nodes (LN) and >0.2 mm but <2 mm.
  S IIA:
  * cancer spread to 1 to 3 LN.
  * tumor <20 mm and spread to the LN.
  * tumor >20 mm but >50 mm
  S IIB:
  * tumor >20 mm but <50 mm and has spread to 1 to 3 LN.
  * tumor >50 mm S IIIA: spread to 4 to 9 LN. S IIIB: tumor spread to the chest wall or caused swelling or ulceration of the breast or is diagnosed as inflammatory breast cancer.
  S IIIC: tumor that has spread to 10 or more LN. S IV: tumor has spread to other organs
  Participants
    Stage I to III | 26
    Stage IV | 22
Prior neo(adjuvant) chemotherapy [Count of Participants; unit: Participants]
  Prior neo(adjuvant) chemotherapy | 23
  Non Prior neo(adjuvant) chemotherapy | 25
Number of disease sites [Count of Participants; unit: Participants]
  1 disease site | 10
  2 disease sites | 18
  3 disease sites or more | 20

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: ORR is the sum of the Complete Responses (CR) and Partial Responses (PR) according to the RECIST criteria, experienced for each patient during treatment (recorded from the start of the treatment until disease progression). Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by CT scan (computed tomography) or MRI (magnetic resonance imaging): Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response Rate (ORR) = CR + PR.
Time Frame: Up to cycle 6 (24 weeks)
Population: 49 patients included but 1 is not considered due to not receive any treatment and died before start
Measure: Count of Participants; unit: Participants
Groups:
- Caelyx,Cyclophosphamide,Trastuzumab: Caelyx (Liposomal Doxorubicin) 50 mg/m2 every 4 weeks for 6 cycles, Cyclophosphamide 600 mg/m2 every 4 weeks for 6 cycles, Trastuzumab weekly for 24 weeks, at dose of 2mg/kg (day 1 loading dose of 4mg/kg)
  Liposomal Doxorubicin
  Cyclophosphamide
  Trastuzumab
Arm/Group | Caelyx,Cyclophosphamide,Trastuzumab
Number analyzed (Participants) | 48
Participants | 33

2. Secondary Outcome: Time to Progression (TTP)
Description: TTP was defined as the time elapsed from first treatment until clinical evidence of disease progression. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: Through study treatment, and follow up period, assessed up to 88 weeks
Population: 49 patients included but 1 is not considered due to not receive any treatment and died before start
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Caelyx,Cyclophosphamide,Trastuzumab
Number analyzed (Participants) | 48
Months | 12 [9 to 15.1]

3. Secondary Outcome: Time to Treatment Failure (TTF)
Description: TTF was defined as the time elapsed from first treatment until patient discontinuation due to toxicity, disease progression, death or withdrawal of consent for any reason, whichever occurred first.
Time Frame: Through study treatment, and follow up period, assessed up to 88 weeks
Population: 49 patients included but 1 is not considered due to not receive any treatment and died before start
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Caelyx,Cyclophosphamide,Trastuzumab
Number analyzed (Participants) | 48
Months | 9.7 [7.9 to 11.4]

4. Secondary Outcome: Response Duration
Description: Response duration was defined as the time elapsed from the first evidence of tumor response (Complete response or Partial Response) until clinical evidence of disease progression or death occurred.
Time Frame: Through study treatment, and follow up period, assessed up to 88 weeks
Population: Patients with Overall Response (see ORR objective)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Caelyx,Cyclophosphamide,Trastuzumab
Number analyzed (Participants) | 33
Months | 9.51 [7.28 to 11.73]

5. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time elapsed from first treatment until death from any cause.
Time Frame: Through study treatment, and follow up period, assessed up to 88 weeks
Population: 49 patients included but 1 is not considered due to not receive any treatment and died before start
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Caelyx,Cyclophosphamide,Trastuzumab
Number analyzed (Participants) | 48
Months | 34.2 [27.2 to 41.2]

ADVERSE EVENTS:
Time Frame: Deaths were assessed for up to 88 weeks. Adverse Events were assessed up to 84 weeks.
Description: 49 patients included but 1 is not considered due to not receive any treatment and died before start
Groups:
- Liposomal Doxorubicin,Cyclophosphamide,Trastuzumab: Liposomal Doxorubicin 50 mg/m2 every 4 weeks for six cycles, Cyclophosphamide 600 mg/m2 every 4 weeks for six cycles, Trastuzumab weekly for 24 weeks, at dose of 2mg/kg (day 1 loading dose of 4mg/kg)
Arm/Group | Liposomal Doxorubicin,Cyclophosphamide,Trastuzumab
All-Cause Mortality (participants affected / at risk) | 2/48
Serious Adverse Events (participants affected / at risk) | 16/48
Other Adverse Events (participants affected / at risk) | 48/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Liposomal Doxorubicin,Cyclophosphamide,Trastuzumab (N=48)
Cerebrovascular ischemia (Nervous system disorders) | 1
Febrile neutropenia grade 3 (Blood and lymphatic system disorders) | 3
Hemorrhage CNS grade 5 (Nervous system disorders) | 1
Infection with normal ANC (skin celluties grade 3) (Skin and subcutaneous tissue disorders) | 1
Acute respiratory insufficiency (Respiratory, thoracic and mediastinal disorders) | 1
Catheter - related infection grade 3 (Infections and infestations) | 1
Holocraneal cephalea (General disorders) | 1
Neutropenia grade 3 (Blood and lymphatic system disorders) | 1
Hemorrhage subarachnoid (Vascular disorders) | 1
Hypersensibility reaction grade 3 (General disorders) | 2
Palmoplantar erythrodysesthesia grade 3, stomatitis grade 3 (General disorders) | 1
Progression disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neutropenia grade 4, fever grade 1, oral mucositis grade 3 (General disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Liposomal Doxorubicin,Cyclophosphamide,Trastuzumab (N=48)
Leukocytes (Blood and lymphatic system disorders) | 1 — Grade 4
Neutrophils / Granulocytes (Blood and lymphatic system disorders) | 5 — Grade 4
Fatigue (General disorders) | 1 — Grade 4
Mucositis / Stomatitis (Gastrointestinal disorders) | 1 — Grade 4
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 2 — Grade 4
Pneumonitis/Pulmonary infiltrates (Reproductive system and breast disorders) | 1 — Grade 5
Leukocytes (Blood and lymphatic system disorders) | 9 — Grade 3
Leukocytes (Blood and lymphatic system disorders) | 10 — Grade 2
Hemoglobin (Blood and lymphatic system disorders) | 10 — Grade 2
Rash: Hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 14 — Grade 3
Mucositis / Stomatitis (Gastrointestinal disorders) | 10 — Grade 3
Lymphopenia (Blood and lymphatic system disorders) | 9 — Grade 2
Lymphopenia (Blood and lymphatic system disorders) | 7 — Grade 3
Neutrophils / Granulocytes (Blood and lymphatic system disorders) | 5 — Grade 3
Neutrophils / Granulocytes (Blood and lymphatic system disorders) | 9 — Grade 2
Left Ventricular systolic dysfunction (Cardiac disorders) | 8 — Grade 2
Fatigue (General disorders) | 16 — Grade 2
Fatigue (General disorders) | 12 — Grade 1
Rash/desquamation (Skin and subcutaneous tissue disorders) | 11 — Grade 2
Rash/desquamation (Skin and subcutaneous tissue disorders) | 8 — Grade 1
Rash: Hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 10 — Grade 2
Rash: Hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 13 — Grade 1
Heartburn/dyspepsia (Gastrointestinal disorders) | 20 — Grade 2
Hemoglobin (Blood and lymphatic system disorders) | 27 — Grade 1
Leukocytes (Blood and lymphatic system disorders) | 14 — Grade 1
Left Ventricular diastolic dysfunction (Cardiac disorders) | 19 — Grade 1
Fever (General disorders) | 9 — Grade 1
Hair loss/alopecia (Skin and subcutaneous tissue disorders) | 12 — Grade 1
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 8 — Grade 1
Anorexia (Gastrointestinal disorders) | 8 — Grade 1
Mucositis / Stomatitis (Gastrointestinal disorders) | 9 — Grade 1
Nausea (Gastrointestinal disorders) | 16 — Grade 1
Infection with normal ANC or G1 or 2 neutrophils (Infections and infestations) | 10 — Grade 2
Alkaline phosphatase (Metabolism and nutrition disorders) | 10 — Grade 1
ALT, SGPT (Metabolism and nutrition disorders) | 20 — Grade 1
AST, SGOT (Metabolism and nutrition disorders) | 18 — Grade 1
Cough (Respiratory, thoracic and mediastinal disorders) | 8 — Grade 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less